CLINICAL TRIAL: NCT06437756
Title: Effects of Theraband Resistance Training on Muscle Strength in Coronary Artery Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/01808 Zunaira Shaukat
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theraband resistance training (Experimental)
  Interventions: Other: Theraband resistance training
- Conventional Resistance Training (Active Comparator)
  Interventions: Other: Conventional Resistance Training

INTERVENTIONS:
Other: Theraband resistance training — Three sessions of 30 minutes each was used to complete the intervention over the course of six weeks (two sets of 12 repetitions). The participants were warmed up by stretching for 10 minutes before each session Participants were advised to take 5 mins rest before moving to next movement if they would feel fatigued after one movement. Thera-Band was utilized in only three different colors for the workouts.
  Arms: Theraband resistance training
Other: Conventional Resistance Training — The intervention was carried out over the course of six weeks in three sessions of 30 minutes each (two sets of 12 repetitions). The participants were warmed up by stretching for 10 minutes before each session. The resistance-training program was performed with Universal weights.
  Arms: Conventional Resistance Training

SUMMARY:
To compare the effects of Theraband Resistance Training with Conventional Resistance Training on muscle strength in coronary artery diseases

ELIGIBILITY:
Inclusion Criteria:

* Participants having a documented diagnosis of CAD, confirmed by a medical professional.
* Individuals with a history of myocardial infarction (heart attack), angina, or evidence of significant coronary artery stenosis.
* Stable CAD who were not experiencing acute coronary events, such as recent heart attacks or unstable angina.
* Patients who were able to perform exercises with TheraBand.
* Reduced muscle strength of upper limb/lower limb

Exclusion Criteria:

* Patients over the age of 75 years.
* Exclude individuals with a recent history of Theraband resistance training.
* Severe cardiovascular complications such as heart failure with reduced ejection fraction, severe arrhythmias, or uncontrolled hypertension.
* Patients with unstable conditions or cardiac episodes.
* Individuals who had undergone major cardiovascular surgery (e.g., coronary artery bypass grafting) within the last six months.
* Ejection fraction < 40%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Hand Held Dynamometer | 6 week
  If testing techniques are consistent, handheld dynamometry is a valid approach to assess the strength state and change in strength status. Hand-held dynamometry can be a reliable assessment technique when practiced by a single experienced tester
Modified BORG Scale | 6 week
  The Modified Borg Dyspnea Scale is numerical rating scale ranging from 0 to 10 and is used to measure dyspnea that patient report during sub-maximal exercise and is regularly administered during six-minute walk test. Changes from the baseline will be measured
Chadler Fatigue Scale | 6 week
  It is a self-administered questionnaire for assessing the degree and severity of fatigue/tiredness in epidemiological populations, both clinical and non-clinical. The Chadler Fatigue Scale (CFS) was originally perceived as comprising two subscales that evaluate fatigue in the physical and mental domains. Items are rated on a 4-point Likert scale (0 = better than usual, 1 = no more than usual, 2 = worse than usual, 3 = much worse than usual), with higher scores indicating greater fatigue. Changes from the baseline are measured
6 Min walk test (Distance in meters) | 6 week
  Changes from the baseline, Body Mass Index can be define as statistical index utilizing an individuals height and weight to give an estimation of muscle versus fat in female and male of all ages. It is determined by taking an individual weight in kilograms, separated by their height in meters squared, or BMI = weight (in kg)/height (in m square).
The 30 Second Sit to Stand Test(30SSST) for lower limb strength | 6 week
  The 30-Second Sit to Stand Test evaluates older people's leg strength and endurance using a foldable chair without arms. Participants stand with feet positioned back from knees, arms crossed, and arms crossed. The examiner counts stand within 30 seconds, determining the score.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Al Nafees Medical Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No